CLINICAL TRIAL: NCT06181448
Title: Real-World Validation of a Prognostic Prediction Model for Patients With Acute Exacerbations of Chronic Liver Disease: A Multi-Site, Prospective Observational Study
Brief Title: Real-World Validation of a Prognostic Prediction Model for Patients With Acute Exacerbations of Chronic Liver Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Hai Li, professor of department of gastroenterological division, Renji Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: Catchlife-predicting
Record Dates: First submitted 2023-12-13; First posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Chronic Liver Disease and Cirrhosis
Keywords: Acute-on-chronic liver failure; Prognostic prediction model; Real-world validation
MeSH Terms: conditions — Fibrosis; Acute-On-Chronic Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hospitalized patients with acute exacerbations of chronic liver disease: 1. Patient data will be collected through a mobile application, providing real-time prognostic scores for patients.
  2. Standary therapy for chronic liver disease with ALI and/or AD

SUMMARY:
Our study is a multi-site, prospective, observational study including patients with acute exacerbations of CLD. Approximately 1500 patients from 24 hospitals in diverse regions in China will be enrolled and followed for 3 months. Data about demographic data, laboratory tests, and clinical manifestations, collected through a mobile application, will inform real-time prognostic scores. The aim of this study is to validate the model's real-world applicability in non-specialist hospital settings.

DETAILED DESCRIPTION:
The study is a multi-site, prospective, observational study conducted in 24 hospitals representing different regions across China. The choice of 24 hospitals was based on their representation of diverse geographical regions across China. These hospitals were selected to ensure a comprehensive validation of the screening model's efficacy in varied healthcare settings. Data will be collected through a mobile application, providing real-time prognostic scores for patients. The study is divided into three parts: patient recruitment, in-hospital follow-up, and post-discharge follow-up . Follow-up will last for 3 months. Endpoints will be considered for all-cause death, survival and liver transplantation. The study is planned to enroll 1500 patients from January 2024 to January 2026.

ELIGIBILITY:
Inclusion Criteria:

* Chronic liver disease with or without cirrhosis, including chronic viral hepatitis, alcoholic liver disease, non-alcoholic fatty liver disease, autoimmune liver disease, metabolic liver disease, chronic drug- induced liver disease and cryptogenic cirrhosis. The duration of underlying non-cirrhotic chronic liver disease should be longer than 6 months.
* Acute exacerbations of chronic liver disease, including acute decompensation (bacterial infection, hepatic encephalopathy, variceal bleeding, ascites and jaundice) in 1 month and liver injury (ALT or AST >3 ULN , or TB>2 ULN) in 1 week.
* Patients are informed of the study purpose and willing to sign the informed consent.

Exclusion Criteria:

* <18 years old or >75 years old
* with malignancy of liver or other organs
* with other serious comorbidities (such as circulatory failure, respiratory failure, chronic kidney disease with end-stage renal failure, stroke within 6 months before admission, severe systemic autoimmune diseases or severe metabolic disease )
* pregnant
* receiving immunosuppressive agents for non-hepatic diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: chronic liver disease patients（with liver dysfunction more than 6 months） with acute liver injury[with ALT>3 ULN),AST>3NL or TB>2 ULN within 1 week before enrollment] or acute decompensation[having ascites, hepatic encephalopathy, bacterial infection ,gastrointestinal bleeding or jaundice(TB > 5ULN)within 1 month before enrollment].
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Short-Term Mortality | 3 months
  All cause mortality within 90 days after admission
Short-Term Liver Transplantation Rate | 3 months
  Liver transplantation rate within 90 days after admission

CONTACTS AND LOCATIONS:
Overall Officials: Hai Li, MD, Study Director — Digestive Department of Renji Hospital,Shanghai Jiao Tong University School of Medicine
Locations (1):
- Renji Hospital,Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided